CLINICAL TRIAL: NCT02069132
Title: Prospective Validation of IWPC Pharmacogenetic Algorithm for Estimating the Appropriate Initial Dose of Warfarin in Elderly People (65 or Older) With Heart Valves Prostheses or Non Valvular Atrial Fibrillation and Comorbidity
Brief Title: Validation of International Warfarin Pharmacogenetics Consortium (IWPC) Algorithm in Elderly Patients With Comorbidity
Acronym: VIALE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Federico II University (Other); University of Salerno (Other)
Responsible Party: Principal Investigator, Ciro Gallo, Professor of Medical Statistics, University of Campania Luigi Vanvitelli
Other Study IDs: VIALE; FARM9JNT9Y (Other Grant/Funding Number: Agenzia Italiana per il Farmaco (AIFA)); 2012-002578-30 (EudraCT Number)
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation; Thrombus Due to Heart Valve Prosthesis
Keywords: Warfarin; International Warfarin Pharmacogenetics Consortium algorithm; Atrial Fibrillation; Heart Valve Prosthesis Implantation; elderly; comorbidity
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Warfarin in elderly with comorbidity: Patients 65 years or older, candidate for therapy with warfarin for non valvular atrial fibrillation or heart valve replacement
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — warfarin treatment will be determined by treating physicians according to in-hospital guidelines, blindly to genotype assessment.

SUMMARY:
The purpose of this study is to validate the International Warfarin Pharmacogenetics Consortium (IWPC) algorithm in a prospective cohort of elderly people (65 years or older) with heart valves and/or nonvalvular atrial fibrillation (AF) and at least one comorbid condition, and to assess the algorithm's prognostic relevance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Patients who initiate warfarin because of non valvular atrial fibrillation or heart valve replacement
* At least one comorbid condition
* At least two other drugs regularly assumed over and above warfarin

Exclusion Criteria:

* Presence of systemic coagulopathies
* Presence of malignancies needing chemotherapy
* Inability or refusal to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: prospective cohort of elderly people (≥65 years) with nonvalvular atrial fibrillation and/or heart valve replacement, with at least one comorbid condition, presenting for warfarin therapy
Sampling Method: Non-Probability Sample
Enrollment: 376 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients whose predicted dose of warfarin is within 20% of the actual stable therapeutic dose. | up to 12 months
  stable warfarin dosing is defined as the mean daily does required to achieve three or more consecutive International Normalized Ratio (INR) measurements within the individual's target range, at the same daily does.

SECONDARY OUTCOMES:
Percentage of patients for whom the predicted dose is at least 20% higher than the actual dose (overestimation) or at least 20% lower than the actual dose (underestimation). | up to 12 months
number of cardiovascular and cerebrovascular events | 12 months
  composite endpoint: death for any cause, hospitalization for cardiovascular and cerebrovascular events, major bleeding or thromboembolism
number of patients with major bleeding events | 12 months
  major bleeding: (i) fatal bleeding; and/or (ii) symptomatic bleeding in a critical area or organ; and/or (iii) bleeding causing a fall in haemoglobin level of ≥2 g/dL or leading to transfusion of two or more units of blood or red cells.
number of thromboembolic event | 12 months
  thromboembolism is defined as occurrence of cerebral infarction, myocardial infarction, peripheral arterial embolism.
number of cardiovascular and cerebrovascular events | 4 weeks
number of patient reported episodes of minor bleeding events | one year
average maintenance dose per patient | 12 months
time to achievement of stable warfarin dosing from initiation | up to 12 months
time to therapeutic INR per patient | up to 12 months
  defined as the time of first achieving INR measurement within the individual's target range, providing that INR is also within the target range at the subsequent clinic visit
percentage time in the therapeutic INR range | up to 3 months
percentage time in the therapeutic INR range | four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Gallo, MD, Study Chair — University of Campania Luigi Vanvitelli; Amelia Filippelli, MD, Principal Investigator — University of Salerno; Marisa De Feo, MD, Principal Investigator — University of Campania Luigi Vanvitelli; Nicola Ferrara, MD, Principal Investigator — Federico II University
Locations (3):
- Italy (3):
  - Second University of Naples, Napoli
  - University of Naples Federico II, Napoli
  - University of Salerno, Salerno